CLINICAL TRIAL: NCT02181569
Title: Sleep Disturbance and Relapse in Individuals With Alcohol Dependence: An Exploratory Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 140143; 14-CC-0143
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2025-11-18

CONDITIONS: Alcoholism
Keywords: Addiction Severity Index; Addiction; Sleep Measures; Sleep Disorders; Natural History
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment seeking participants with alcohol dependence: Treatment seeking individuals with alcohol dependence who are admitted into a 28-day inpatient treatment program.

SUMMARY:
Despite research establishing the relationship between sleep disturbances and alcohol use, there is no clear understanding or model for what occurs once individuals who seek inpatient alcoholism treatment are discharged from rehabilitation facilities and attempt to integrate back into their homes and communities. The purpose of this investigation will be to characterize sleep patterns, perceptions, and beliefs throughout the process of alcohol rehabilitation. The misuse of alcohol is a global public health concern that compromises both individual and societal wellbeing, resulting in an estimated 2.5 million deaths annually. The National Institute on Alcohol Abuse and Alcoholism (NIAAA) distinguishes alcoholism by craving, loss of control, physical dependence, and tolerance (NIAAA, Alcohol Use Disorders). The relationship between alcohol use and sleep disturbances is complex and bidirectional, but sleep disturbances are common among alcoholics during phases of drinking, withdrawal, and abstinence. Outcome expectancies, behavioral capability, and self-efficacy beliefs are central constructs in the Social Cognitive Theory and will be measured directly in this study using both quantitative and qualitative methods. A mixed methods approach will be used to study the following aims: a) to assess individuals' perceptions of and experiences with sleep during alcohol rehabilitation, b) to describe sleep patterns, perceptions, and beliefs among alcohol-dependent individuals throughout the transition from a clinical research facility providing rehabilitation treatment back to the community, c) to assess whether sleep-related beliefs and/or behavior of individuals are predictive of sleep quality or relapse to drinking, and d) to assess whether sleep quality predicts relapse. Adult research participants admitted to the inpatient behavioral health unit and enrolled on to the NIAAA intramural study NCT 0010693: Assessment and Treatment of People with Alcohol Drinking Problems will be recruited for participation in this study (n=215). Sleep quality and duration will be quantitatively assessed approximately one week prior to discharge from the inpatient facility and again 4-6 weeks post-discharge. A sub-set of participants will be asked to wear actiwatches (accelerometers) to provide objective data on sleep throughout the transition from inpatient to outpatient. In addition to quantitative measures, qualitative semi-structured interviews will be conducted with a subset of 25 participants (to reach 25 completed cases) within a week of the scheduled discharge date and again four to six weeks post-discharge to assess perceptions of sleep during recovery. The proposed study will fill a gap in the literature by characterizing sleep throughout the rehabilitation process and ongoing maintenance of abstinence.

DETAILED DESCRIPTION:
Despite research establishing the relationship between sleep disturbances and alcohol use, there is no clear understanding or model for what occurs once individuals who seek inpatient alcoholism treatment are discharged from rehabilitation facilities and attempt to integrate back into their homes and communities. The purpose of this investigation will be to characterize sleep patterns, perceptions, and beliefs throughout the process of alcohol rehabilitation. The misuse of alcohol is a global public health concern that compromises both individual and societal wellbeing, resulting in an estimated 2.5 million deaths annually. The National Institute on Alcohol Abuse and Alcoholism (NIAAA) distinguishes alcoholism by craving, loss of control, physical dependence, and tolerance (NIAAA, Alcohol Use Disorders). The relationship between alcohol use and sleep disturbances is complex and bidirectional, but sleep disturbances are common among alcoholics during phases of drinking, withdrawal, and abstinence. Outcome expectancies, behavioral capability, and self-efficacy beliefs are central constructs in the Social Cognitive Theory and will be measured directly in this study using both quantitative and qualitative methods. A mixed methods approach will be used to study the following aims: a) to assess individuals' perceptions of and experiences with sleep during alcohol rehabilitation, b) to describe sleep patterns, perceptions, and beliefs among alcohol-dependent individuals throughout the transition from a clinical research facility providing rehabilitation treatment back to the community, c) to assess whether sleep-related beliefs and/or behavior of individuals are predictive of sleep quality or relapse to drinking, and d) to assess whether sleep quality predicts relapse. Adult research participants admitted to the inpatient behavioral health unit and enrolled on to the NIAAA intramural study NCT 0010693: Assessment and Treatment of People with Alcohol Drinking Problems will be recruited for participation in this study (n=215). Sleep quality and duration will be quantitatively assessed approximately one week prior to discharge from the inpatient facility and again 4-6 weeks post-discharge. A sub-set of participants will be asked to wear actiwatches (accelerometers) to provide objective data on sleep throughout the transition from inpatient to outpatient. In addition to quantitative measures, qualitative semi-structured interviews will be conducted with a subset of 25 participants (to reach 25 completed cases) within a week of the scheduled discharge date and again four to six weeks post-discharge to assess perceptions of sleep during recovery. The proposed study will fill a gap in the literature by characterizing sleep throughout the rehabilitation process and ongoing maintenance of abstinence.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible for this study if they are:

* 18 years of age or older,
* Enrolled on the screening, assessment and treatment protocol (14-AA-0181)
* Have been an inpatient for 21 days or more preceding discharge,
* Not enrolled onto a pharmacologic intervention study,
* Able to understand the study, and
* Willing to return to the Clinical Center 4-6 weeks after being discharged from inpatient treatment for a follow-up visit.

EXCLUSION CRITERIA:

Participants will be ineligible for this study if they are:

* Less than 18 years of age,
* Unable to understand the purpose of the study,
* Unable to provide informed consent,
* Unable to follow the study design, or
* Unable or unwilling to return to the Clinical Center 4-6 weeks after being discharged from inpatient treatment for a follow-up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment seeking individuals with alcohol dependence who are admitted into a 28-day inpatient treatment program.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
PSQI | Day 2 of inpatient admission, within 7 days of discharge, and 4-6 weeks after discharge
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item, self-rated questionnaire used to measure sleep quality and disturbances over a one-month (30 days) time interval. Nineteen individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A global summation score of five or higher is indicative of poor sleep quality (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). The PSQI has been validated in populations with insomnia and other sleep disorders, with psychiatric patients, and in normal populations (Backhaus, Junghanns, Broocks, Riemann, & Hohagen, 2002; Doi, Minowa, Uchiyama, Okawa, Kim, Shibui, & Kamei, 2000).

SECONDARY OUTCOMES:
TLFB | Day 13 and 4-6 weeks after discharge
  The TLFB collects drinking information using personal historical events recounted over a fixed time period (Sobell & Sobell, 1992). It is a standard assessment for measuring alcohol drinking patterns and quantification in treatment programs. The number of items corresponds to the number of days of interest, typically 90, which usually takes about 30 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Barb-Smith, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-CC-0143.html